CLINICAL TRIAL: NCT00695773
Title: Laparoscopic Vs. Open Prostatectomy Outcomes
Status: Terminated | Type: Observational
Why Stopped: Insufficient findings for data analysis
Sponsor: Lahey Clinic (Other)
Responsible Party: John A. Libertino, M.D., Lahey Clinic, Inc.
Other Study IDs: 2006-014
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Prostate Cancer Surgery
Keywords: Prostate Cancer Surgery; Laparoscopic surgery for Prostate Cancer; Prostatectomy; Urologic Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is aimed at discovering the differences in outcomes, regarding quality of life issues(continence, impotence) of patients who have had either laparoscopic or open surgical technique for prostate cancer.

DETAILED DESCRIPTION:
This study is a post surgical, data collection effort in order to gather definitive, Quality of Life(continence, impotence) information regarding the outcomes of patients who have undergone either Laparoscopic vs. Prostatectomy surgeries for Prostate Cancer. As part of the study, 200 subject's medical records will be retrospectively reviewed and 100 current subjects will be prospectively contacted. The information collected may benefit patients who undergo a prostatectomy

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone a prostatectomy

Exclusion Criteria:

* none

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A Lahey Clinic IRB approved database and current clinic population of patients having a laparascopic or open prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2006-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The post-surgical questionnaire information collected will be used to determine any benefits to future patients who are to undergo a prostatectomy | Post Surgical

CONTACTS AND LOCATIONS:
Overall Officials: John A. Libertino, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States